CLINICAL TRIAL: NCT03440866
Title: Comparison of the Effectiveness of Treatment With Mifepristone and Misoprostol at the Same Time Compared to the Administration of Drugs at a 48-hour Interval for Medical Abortion in Young Pregnancy - A Prospective Randomized Controlled Trial.
Brief Title: Comparison of the Effectiveness of Treatment With Mifepristone and Misoprostol at the Same Time Compared to the Administration of Drugs at a 48-hour Interval for Medical Abortion.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2-17 EMC
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Early Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Administration of drugs concomitantly.
  Interventions: Drug: Administration of drugs concomitantly.
- Control (No Intervention): Administration of oral Mifepristone 600 mg and after interval of 48 hours administration of oral Misoprostol 400 mcg.

INTERVENTIONS:
Drug: Administration of drugs concomitantly. — Administration of oral Mifepristone 600 mg and oral Misoprostol 400 mcg concomitantly.
  Other Names: no interval
  Arms: Intervention

SUMMARY:
Medical termination of pregnancy is a common and safe alternative to surgical termination of pregnancy(8). The current protocol in the investigators unit includes oral administration of Mifepristone 600 mg and oral Misoprostol 400 mcg in a time interval of 48 hours. There is little data to compare the efficacy of concomitant administration of both drugs and different time intervals.

This study evaluates the success rate and side effects of medical termination of pregnancy while both drugs are administrated concomitantly in comparison to interval of 48 hours between the drugs.

DETAILED DESCRIPTION:
Medical termination of pregnancy is a common and safe alternative to surgical termination of pregnancy(8). According to the original protocol ,the administration of oral Mifepristone 600 mg is followed by oral Misoprostol 400 mcg in an interval of 36 to 48 hours. Shortening this time interval may convince patients to avoid surgical termination of pregnancy, enhance patient's compliance to treatment and even be more economically.

The current protocol in the investigators unit includes oral administration of Mifepristone 600 mg and oral Misoprostol 400 mcg in a time interval of 48 hours. The patients are recommended to have an ultrasound examination after 2 to 3 weeks. There is little data to compare the efficacy of concomitant administration of both drugs according to the dosage of this protocol and different time intervals.

This study evaluates the success rate and side effects of medical termination of pregnancy while both drugs are administrated concomitantly in comparison to interval of 48 hours between the drugs.

Participants in the study group will be given both drugs at the same time while participants in the control group will be given Mifepristone and Misoprostol in an interval of 48 hours.

The investigators hypothesis is that administration of both drugs concomitantly will not change significantly the success rate of the procedure and will not enhance the side effects.

ELIGIBILITY:
Inclusion Criteria:

* intrauterine singleton pregnancy of less than 49 days, reassured by ultrasound examination
* patient who desire to terminate their pregnancy and have approval of the committee for termination of pregnancy
* patient who gave their consent to have a surgical abortion eventual if needed

Exclusion Criteria:

* contraindication to Mifepristone or Misoprostol
* suspected ectopic pregnancy
* systemic treatment with steroids
* adrenal insufficiency
* heart and blood vessels disease
* coagulopathy or use of anti-thrombotic agents
* uncontrolled asthma
* liver or kidney insufficiency
* anorexia
* intrauterine device
* breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of complete abortion | two weeks
  Success rate of complete abortion without any other surgical intervention

SECONDARY OUTCOMES:
Bleeding amount | two weeks
  Assessment of bleeding amount and duration by the patient (maximum amount of pads per day) and Hemoglobin level before and two weeks after the procedure
Self reported pain intensity after two weeks | two weeks
  Visual analogue scale pain severity with scale from 0 to 10, with score 10 representing the maximum level of pain during those two weeks.
patient's satisfaction | two weeks
  Post operative women's satisfaction with scale from 0 to 10, with score 10 representing the maximum level of satisfaction. the patient will be asked if she will select this method next time if necessary

CONTACTS AND LOCATIONS:
Overall Officials: meirav braverman, MD, Principal Investigator — HaEmek Medical Center, Afula, Israel
Locations (1):
- HaEmek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Creinin MD, Schreiber CA, Bednarek P, Lintu H, Wagner MS, Meyn LA; Medical Abortion at the Same Time (MAST) Study Trial Group. Mifepristone and misoprostol administered simultaneously versus 24 hours apart for abortion: a randomized controlled trial. Obstet Gynecol. 2007 Apr;109(4):885-94. doi: 10.1097/01.AOG.0000258298.35143.d2. PMID 17400850
- [Result] Termination of pregnancy with reduced doses of mifepristone. World Health Organisation Task Force on Post-ovulatory Methods of Fertility Regulation. BMJ. 1993 Aug 28;307(6903):532-7. doi: 10.1136/bmj.307.6903.532. PMID 8400972
- [Result] McKinley C, Thong KJ, Baird DT. The effect of dose of mifepristone and gestation on the efficacy of medical abortion with mifepristone and misoprostol. Hum Reprod. 1993 Sep;8(9):1502-5. doi: 10.1093/oxfordjournals.humrep.a138287. PMID 8253942
- [Result] Creinin MD, Schwartz JL, Pymar HC, Fink W. Efficacy of mifepristone followed on the same day by misoprostol for early termination of pregnancy: report of a randomised trial. BJOG. 2001 May;108(5):469-73. doi: 10.1111/j.1471-0528.2001.00117.x. PMID 11368131
- [Result] World Health Organisation Task Force on Post-ovulatory Methods of Fertility Regulation; Special Programme of Research, Development and Research Training; World Health Organisation. Comparison of two doses of mifepristone in combination with misoprostol for early medical abortion: a randomised trial. BJOG. 2000 Apr;107(4):524-30. doi: 10.1111/j.1471-0528.2000.tb13273.x. PMID 10759273
- [Result] Creinin MD, Fox MC, Teal S, Chen A, Schaff EA, Meyn LA; MOD Study Trial Group. A randomized comparison of misoprostol 6 to 8 hours versus 24 hours after mifepristone for abortion. Obstet Gynecol. 2004 May;103(5 Pt 1):851-9. doi: 10.1097/01.AOG.0000124271.23499.84. PMID 15121556
- [Result] von Hertzen H, Piaggio G, Wojdyla D, Marions L, My Huong NT, Tang OS, Fang AH, Wu SC, Kalmar L, Mittal S, Erdenetungalag R, Horga M, Pretnar-Darovec A, Kapamadzija A, Dickson K, Anh ND, Tai NV, Tuyet HT, Peregoudov A; WHO Research Group on Post-ovulatory Methods of Fertility Regulation. Two mifepristone doses and two intervals of misoprostol administration for termination of early pregnancy: a randomised factorial controlled equivalence trial. BJOG. 2009 Feb;116(3):381-9. doi: 10.1111/j.1471-0528.2008.02034.x. PMID 19187370
- [Result] Garg G, Takkar N, Sehgal A. Buccal versus vaginal misoprostol administration for the induction of first and second trimester abortions. J Obstet Gynaecol India. 2015 Apr;65(2):111-6. doi: 10.1007/s13224-014-0605-5. Epub 2014 Oct 31. PMID 25883442
- [Result] Murthy AS, Creinin MD, Harwood B, Schreiber C. A pilot study of mifepristone and misoprostol administered at the same time for abortion up to 49 days gestation. Contraception. 2005 May;71(5):333-6. doi: 10.1016/j.contraception.2004.10.006. PMID 15854632
- [Result] Goel A, Mittal S, Taneja BK, Singal N, Attri S. Simultaneous administration of mifepristone and misoprostol for early termination of pregnancy: a randomized controlled trial. Arch Gynecol Obstet. 2011 Jun;283(6):1409-13. doi: 10.1007/s00404-011-1881-2. Epub 2011 Mar 23. PMID 21431329
- [Result] Schaff E. Evidence for shortening the time interval of prostaglandin after mifepristone for medical abortion. Contraception. 2006 Jul;74(1):42-4. doi: 10.1016/j.contraception.2006.03.014. Epub 2006 May 12. PMID 16781259
- [Result] Schaff EA, Fielding SL, Westhoff C. Randomized trial of oral versus vaginal misoprostol at one day after mifepristone for early medical abortion. Contraception. 2001 Aug;64(2):81-5. doi: 10.1016/s0010-7824(01)00229-3. PMID 11704083
- [Result] Wedisinghe L, Elsandabesee D. Flexible mifepristone and misoprostol administration interval for first-trimester medical termination. Contraception. 2010 Apr;81(4):269-74. doi: 10.1016/j.contraception.2009.09.007. Epub 2009 Oct 29. PMID 20227541
- [Derived] Braverman M, Dayan-Schwartz A, Ben-David Y, Kachta O, Zafran N. Early Pregnancy Termination with Mifepristone and Misoprostol: Concurrent vs. 48-Hour Interval Administration in a Randomized Controlled Trial. J Clin Med. 2025 Oct 27;14(21):7616. doi: 10.3390/jcm14217616. PMID 41227012